CLINICAL TRIAL: NCT04732299
Title: Staging Diagnosis and Prognosis of Lower Extremity Deep Venous Thrombosis Based on Magnetic Resonance Imaging: a Prospective Study
Brief Title: Staging and Prognosis of Deep Venous Thrombosis of Lower Extremities
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2020-014
Record Dates: First submitted 2021-01-28; First posted 2021-02-01 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Venous Thrombosis
Keywords: MRI, Venous Thrombosis, Staging, Prognosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acute thrombus group: Within 14 days after onset
  Interventions: Other: MRI examination
- Subacute thrombus group: During 15-30 days after onset
  Interventions: Other: MRI examination
- Chronic thrombosis group: More than 15-30 days after onset
  Interventions: Other: MRI examination

INTERVENTIONS:
Other: MRI examination — Magnetic resonance thrombography is used to determine the location of thrombus, quantify the thrombus and determine its stage.

SUMMARY:
Deep venous thrombosis (DVT) is a venous reflux disorder caused by abnormal coagulation of blood in the deep vein, which usually occurs in the lower extremities. After thrombosis, venous valve function is often destroyed, causing lower limb swelling, ulcers and other congestive diseases, affecting the quality of life of patients; thrombus shedding is also easy to cause pulmonary embolism, serious cases can lead to sudden death. Therefore, the accurate diagnosis and curative effect evaluation of DVT are of great significance to the prognosis of patients. At present, the treatment of DVT includes systematic thrombolysis and catheter contact thrombolysis, among which oral drug thrombolysis has certain advantages in clinical application. However, in the process of thrombosis, the composition of thrombus is different in different periods, thus, defining the staging of thrombus plays an important role in the decision-making of drug treatment. In view of the high resolution of magnetic resonance imaging of soft tissue, thrombus can be directly imaged. Therefore, this project will take the staging diagnosis of deep venous thrombosis as the starting point. Through the development of magnetic resonance imaging, this paper tries to solve the problem of evaluating the therapeutic effect of deep venous thrombosis in clinic.

DETAILED DESCRIPTION:
Deep venous thrombosis (DVT) is a venous reflux disorder caused by abnormal blood coagulation in the deep vein, which usually occurs in the lower extremities. DVT is common in patients with limb immobilization (such as after major orthopedic surgery), severe trauma, tumor, coma or long-term bedridden patients. After thrombosis, venous valve function is often destroyed, causing lower limb swelling, ulcers and other congestive diseases, affecting the quality of life of patients; thrombus shedding is also easy to cause pulmonary embolism, serious cases can lead to sudden death.

In the process of thrombosis, the components of thrombus are different in different stages. in the acute stage of thrombosis, the consumption of blood fibroses is less, mainly in the thrombolytic therapy of activating plasminogen; in the subacute and chronic phase of thrombosis, the consumption of fibrinolytic enzyme is more, anticoagulant therapy is needed to prolong the clotting time. Therefore, defining the staging of thrombus is the key to make a reasonable treatment plan and improve the therapeutic effect of DVT. The guidelines recommend that for patients with moderate or high likelihood of DVT, if two consecutive ultrasound examinations are negative, further X-ray venography, CT venography or magnetic resonance venous thrombosis direct imaging are recommended. Among them, magnetic resonance thrombus direct imaging depends on the content of methemoglobin in the body and will not produce radiation to the human body. it can not only accurately judge the thrombus in the pelvic and inferior vena cava, but also show the details of the changes in the vein wall or lumen. Therefore, magnetic resonance thrombus direct imaging has a certain potential in the differential diagnosis of acute, subacute and old thrombus. In this study, we will use magnetic resonance thrombus direct imaging to stage and judge the efficacy of drug treatment, in order to provide help for clinic.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* Suspected deep venous thrombosis of lower extremities
* No treatment related to deep venous thrombosis of lower extremities

Exclusion Criteria:

* Contraindication of magnetic resonance imaging
* Previous history of deep venous thrombosis
* History of allergy to magnetic resonance contrast agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The people included in this study are patients suspected of deep venous thrombosis of lower extremities for the first time and should be older than 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-06-15 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Thrombus-muscle signal-to-noise ratio | The interval between two MRI examinations per patient is 3 months.
  Quantitative analysis of thrombus was performed by magnetic resonance thrombography for the first time, and the curative effect was evaluated again 3 months after clinical treatment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dronkers CE, Sramek A, Huisman MV, Klok FA. Accurate diagnosis of iliac vein thrombosis in pregnancy with magnetic resonance direct thrombus imaging (MRDTI). BMJ Case Rep. 2016 Dec 13;2016:bcr2016218091. doi: 10.1136/bcr-2016-218091. PMID 27965311
- [Background] Karande GY, Hedgire SS, Sanchez Y, Baliyan V, Mishra V, Ganguli S, Prabhakar AM. Advanced imaging in acute and chronic deep vein thrombosis. Cardiovasc Diagn Ther. 2016 Dec;6(6):493-507. doi: 10.21037/cdt.2016.12.06. PMID 28123971
- [Background] Mendichovszky IA, Priest AN, Bowden DJ, Hunter S, Joubert I, Hilborne S, Graves MJ, Baglin T, Lomas DJ. Combined MR direct thrombus imaging and non-contrast magnetic resonance venography reveal the evolution of deep vein thrombosis: a feasibility study. Eur Radiol. 2017 Jun;27(6):2326-2332. doi: 10.1007/s00330-016-4555-4. Epub 2016 Aug 30. PMID 27578046
- [Background] Xie G, Chen H, He X, Liang J, Deng W, He Z, Ye Y, Yang Q, Bi X, Liu X, Li D, Fan Z. Black-blood thrombus imaging (BTI): a contrast-free cardiovascular magnetic resonance approach for the diagnosis of non-acute deep vein thrombosis. J Cardiovasc Magn Reson. 2017 Jan 18;19(1):4. doi: 10.1186/s12968-016-0320-8. PMID 28095878
- [Background] Chen H, He X, Xie G, Liang J, Ye Y, Deng W, He Z, Liu D, Li D, Liu X, Fan Z. Cardiovascular magnetic resonance black-blood thrombus imaging for the diagnosis of acute deep vein thrombosis at 1.5 Tesla. J Cardiovasc Magn Reson. 2018 Jun 25;20(1):42. doi: 10.1186/s12968-018-0459-6. PMID 29936910
- [Background] Zhuang G, Tang C, He X, Liang J, He Z, Ye Y, Deng W, Liu D, Chen H. DANTE-SPACE: a new technical tool for DVT on 1.5T MRI. Int J Cardiovasc Imaging. 2019 Dec;35(12):2231-2237. doi: 10.1007/s10554-019-01675-w. Epub 2019 Aug 24. PMID 31446527